CLINICAL TRIAL: NCT03744403
Title: A Phase I, Open-Label, Multiple-Dose, Dose-Escalation Study of an Anti-PD-L1 Monoclonal Antibody CS1001 in Subjects with Advanced Solid Tumors
Brief Title: A Study of CS1001 in Subjects with Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CStone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS1001-102
Record Dates: First submitted 2018-11-14; First posted 2018-11-16 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2022-02

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CS1001 monoclonal antibody (Experimental)
  Interventions: Drug: CS1001

INTERVENTIONS:
Drug: CS1001 — In the dose-escalation part, the dose levels will be escalated following a modified 3+3 dose escalation scheme. In the dose-expansion part, both dose levels will be expanded.

SUMMARY:
This is a phase I, open-label, multiple-dose, dose-escalation study to evaluate the safety, tolerability, pharmacokinetics and anti-tumor activity of CS1001 in subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with metastatic or locally advanced unresectable solid tumor, who progressed following treatment with all available standard therapy, or for whom treatment is not available, not tolerated or refused.
2. ECOG performance status of 0 or 1.
3. Subjects must have at least one measurable lesion.
4. Patients with life expectancy ≥ 3 months.
5. Subject must have adequate organ function.
6. Fertile men and women of childbearing potential must agree to use an effective method of birth control from providing signed consent and for 180 days after last study drug administration.

Exclusion Criteria:

1. Known brain metastasis or other CNS metastasis that is either symptomatic or untreated.
2. Subjects with active autoimmune diseases or history of autoimmune diseases should be excluded.
3. Patients who have received prior therapies targeting PD-1, PD-L1, or CTLA-4.
4. Known history of HIV infection.
5. Subjects with active Hepatitis B or C infection.
6. Any unresolved CTCAE Grade ≥ 2 toxicities from prior anti-cancer therapy with the exception of vitiligo, alopecia.
7. Patients who have serious hypersensitive reaction to monoclonal antibodies, and have history of uncontrolled allergic asthma.
8. Known history of alcoholism or drugs abuse.
9. Subjects who received organ transplantation.
10. Known psychiatric disorders that would interfere with cooperation with the requirements of the trial.
11. Female subjects who are pregnant or breast-feeding; Male or female subjects of childbearing potential who refuse to use an effective method of birth control.

For more information regarding trial participation, please contact at cstonera@cstonepharma.com

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2021-07-21 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | From first dose to 90 days after last dose of CS1001, up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- NEXT Oncology, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No